CLINICAL TRIAL: NCT03050567
Title: Reproducibility Study of Transcranial Doppler Microembolic Signals Detection in the Middle Cerebral Artery
Brief Title: Reproducibility Study of Transcranial Doppler
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC16131
Record Dates: First submitted 2016-11-16; First posted 2017-02-13 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: Microemboli
MeSH Terms: conditions — Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers with no previous history of cerebrovascular disease and aged over 18 years old.
  Interventions: Diagnostic Test: Transcranial Doppler Ultrasound
- Subjects with symptomatic carotid artery stenosis: Patients with symptomatic cerebrovascular event (stroke, transient ischaemic attack or amaurosis fugax) and image confirmed carotid artery stenosis of >30%. This will include patients scheduled for carotid endarterectomy (>50% for men and >70% for women, by North American Symptomatic Carotid Endarterectomy Trial criteria) or treated conservatively with an optimal medical therapy (if patient declined surgical intervention or is outside surgical criteria for carotid endarterectomy).
  Interventions: Diagnostic Test: Transcranial Doppler Ultrasound

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler Ultrasound — Transcranial Doppler will be performed on the symptomatic (ipsilateral to an index event) middle cerebral artery in a quiet temperature controlled room. The middle cerebral artery will be identified through the temporal window in a supine position with a flow direction towards the probe. The subject will have a head frame (Marc 600 Spencer Technologies, USA) fitted to reduce motion and to secure a constant angle of the middle cerebral artery insonation depth at 50-60 mm from the skull surface. All recordings will be made using the ST3 Transcranial Doppler Ultrasound System (Spencer Technologies, USA) with a 2-MHz transducer for 1 hour. Emboli will be detected by listening for their characteristic short audible sound (range 10-100 ms, intensity threshold above 7 dB) and spectral appearance using the International Consensus Group microembolus identification criteria and an automated Embolus Detection Software (Spencer Technologies, USA).

SUMMARY:
Hardening of the neck vessels (carotid arteries) caused by fatty deposits called 'plaques' is a common cause of strokes. Over time plaques can burst or may lead to a severe narrowing (stenosis) of the neck artery. When plaques burst, small clots or fatty particles (called microemboli) break off, block brain vessels and lead to a stroke. Researchers have an incomplete understanding of the processes that cause hardening of the arteries, development of small clots and are unable to predict who will have a stroke. At present, the only ultrasound scan that evaluates circulation in the head and detects these small clots is called the Transcranial Doppler ultrasound. The aim of the study is to test this simple ultrasound technique to see if it can detect signals that may correspond to these small clots or fatty particles. The other objective is to see how repeatable the ultrasound technique is. This may help to identify patients with hardened neck arteries who are at higher risk of a recurrent stroke. This could also potentially improve patients selection to a targeted surgical or future novel pharmacological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with no previous history of cerebrovascular disease and aged over 18 years old.
* Patients with symptomatic cerebrovascular event (stroke, transient ischaemic attack or amaurosis fugax) and image confirmed carotid artery stenosis of >30%. This will include patients scheduled for carotid endarterectomy (>50% for men and >70% for women, by North American Symptomatic Carotid Endarterectomy Trial criteria) or treated conservatively with an optimal medical therapy (if patient declined surgical intervention or is outside surgical criteria for carotid endarterectomy).

Exclusion Criteria:

* Subjects unable to comply with the study procedures such as a severe disabling stroke.
* Inadequate temporal window for Transcranial Doppler assessment.
* Adults with incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two cohorts of subjects including healthy volunteers and those with symptomatic carotid artery stenosis will be recruited in different ways. All subjects will undergo basic clinical evaluation prior to participation. In the second cohort, this will include assessment of relevant carotid artery and brain imaging investigations as well.
  Healthy volunteers will be recruited from the Centre for Cardiovascular Science at Edinburgh University by the Primary Investigator (PI).
  Patients with evidence of an acute neurovascular event (stroke, transient ischaemic attach and retinal ischaemia) due to a symptomatic carotid artery stenosis will be recruited from the acute TIA/Stroke clinics and inpatients at Edinburgh Royal Infirmary by the responsible Consultant Neurologist or Stroke Physician. Once eligible patients are identified at this point PI will recruit subjects into the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Presence of microembolic signals in the Middle Cerebral Artery. | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Kaczynski J, Home R, Shields K, Walters M, Whiteley W, Wardlaw J, Newby DE. Reproducibility of Transcranial Doppler ultrasound in the middle cerebral artery. Cardiovasc Ultrasound. 2018 Sep 11;16(1):15. doi: 10.1186/s12947-018-0133-z. PMID 30200977